CLINICAL TRIAL: NCT03515343
Title: Optivista : I-SCAN OE for Optical Diagnosis of Small Colon Polyps
Acronym: Optivista
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Pentax Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 17.135
Record Dates: First submitted 2018-03-15; First posted 2018-05-03 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2018-03

CONDITIONS: Colo-rectal Cancer; Polyps of Colon
Keywords: Cancer prevention; Endoscopy; Gastroenterology
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Biopsy of colorectal polyps detected during the observed colonoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Optical diagnosis with Optivista: Participants for which the optical diagnosis of detected colorectal polyps will be done with the new technique Pentax Optivista.
  Interventions: Diagnostic Test: Screening colonoscopy according to resect-and-discard strategy
- Optical diagnosis with iScan: Participants for which the optical diagnosis of detected colorectal polyps will be done with the oldest technique Pentax iScan.
  Interventions: Diagnostic Test: Screening colonoscopy according to resect-and-discard strategy

INTERVENTIONS:
Diagnostic Test: Screening colonoscopy according to resect-and-discard strategy — This strategy uses image enhancing techniques and optical diagnosis instead of histopathology assessment with 2 Pentax optical imaging systems (either Optivista or iScan).

SUMMARY:
This prospective randomized clinical trial aims to evaluate the new Optivista system compared to the iScan for his optical diagnosis and interval agreement monitoring with pathology. The Participants will be randomized to be diagnosed by either Optivista or Pentax iScan, and all polyps detected during the procedure, their size, location and morphology will be recorded according to the Paris classification after which all polyps will be resected per standard practices and sent for histopathologic evaluation. Further optical assessments will be performed for all polyps of 1-10 mm in size (WASP, NICE, SANO and SIMPLE classification) after with an analysis of comparison between optical diagnosis and pathology results will be performed.

DETAILED DESCRIPTION:
The benefit of colonoscopy screening is based on the detection and removal of polyps neoplastic. However, the vast majority of found polyps do not harbor any risk of non-cancer neoplastic. The resection evaluation and histopathology of these polyps are associated with costs while the contribution to cancer prevention is limited. A new technique (Pentax Optivista) based on visual diagnosis of polyps has been introduced to reduce the costs associated with over-screening, and seems to be more efficient than the Pentax iScan technique.

This research project aims to evaluate the new Optivista system compared to the iScan for his optical biopsy performance and interval agreement monitoring with pathology.

This is a prospective clinical trial for which participants are recruited directly from the colonoscopy clinic. The Participants will be randomized to be diagnosed by either Optivista or Pentax iScan. Endoscope withdrawal will be done in iScan 1 mode for patients randomized to iSan and in Optivista OE2 mode for patients randomized to Optivista.

For all polyps detected during the procedure, their size, location and morphology will be recorded according to the Paris classification after which all polyps will be resected per standard practices and sent for histopathologic evaluation.

Polyps that are between 1-10mm in size (diminutive and small polyps), there will be further assessed according to WASP, NICE, SANO and SIMPLE classifications using white light imaging and using an image-enhancing endoscopy technology that enhances visualisation of the polyp surface and vascular patterns.

Concordance between optical diagnosis and pathology monitoring according to recommendations will be presented as proportions with a 95% CI. The features optical polyp diagnostic test for overall diminutive (1-5mm) polyps and by location in the colon (proximal, distal, colon and rectosigmoid segments) will be presented. For outcome measures secondary factors, including factors that may influence the optical diagnosis, proportional estimates with a 95% confidence interval (CI) will be presented. Concordance between strategies is examined using a marginal homogeneity test (Stuart-Maxwell test). For the comparison of proportions, a chi square test or a Fisher's exact two-sided test will be used, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Aged 45 to 80 years
* Indication for full colonoscopy

Exclusion Criteria:

* Known inflammatory bowel disease
* Active colitis
* Coagulopathy
* Familial polyposis syndrome
* Poor general health defined as an ASA class > 3
* Emergency colonoscopies

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited at the endoscopy unit at the CHUM, before undergoing an elective colonoscopy.
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Concordance of Optical diagnosis with the pathology based reference standard | 12 months
  The Optical diagnosis of polyps using Optivista or iScan will be compared with the pathology based reference standard.
Rate of polyps detected of both of the technologies (Optivista and iScan) for Optical diagnosis | 12 months

SECONDARY OUTCOMES:
Negative predictive value of rectosigmoid neoplastic polyps. | 12 months
  Secondary outcomes and data collection include test characteristics, particularly the negative predictive value of rectosigmoid neoplastic polyps.
Concordance of biopsies with WASP classification | 12 months
  Verification of concordance (yes/no) between histopathological results (biopsies) and WASP classification for polyps up to 10mm in size in conjunction with iScan and Optivista (depending on randomization).
Concordance of biopsies and SIMPLE classification | 12 months
  Verification of concordance (yes/no) between histopathological results (biopsies) and SIMPLE classification for polyps up to 10mm in size in conjunction with iScan and Optivista (depending on randomization).
Concordance of biopsies and SANO classification | 12 months
  Verification of concordance (yes/no) between histopathological results (biopsies) and SANO classification for polyps up to 10mm in size in conjunction with iScan and Optivista (depending on randomization).
Concordance of biopsies and NICE classification | 12 months
  Verification of concordance (yes/no) between histopathological results (biopsies) and NICE classification for polyps up to 10mm in size in conjunction with iScan and Optivista (depending on randomization).
Surveillance recommendation following the colonoscopy | 12 months
  The proportion of patients for whom an immediate surveillance recommendation following the colonoscopy can be directly provided for each approach and how often histopathology polyp examination would have been avoided when using each strategy will be examined.
Evaluate Polyp-Based Resect and Discard model | 12 months
  Surveillance interval agreement of the PBRD strategy compared with pathology-based management according to the 2020 USMSTF guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Montréal, Research Center (CRCHUM)
Locations (1):
- Centre Hospitalier Universitaire de Montréal (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Djinbachian R, Marchand E, Pohl H, Aguilera-Fish A, Bouin M, Deslandres E, Weber A, Bouchard S, Panzini B, von Renteln D. Optical diagnosis of colorectal polyps: a randomized controlled trial comparing endoscopic image-enhancing modalities. Gastrointest Endosc. 2021 Mar;93(3):712-719.e1. doi: 10.1016/j.gie.2020.11.023. Epub 2020 Dec 2. PMID 33275913